CLINICAL TRIAL: NCT07249554
Title: Preliminary Safety and Efficacy of Semaglutide and Naltrexone Combination Therapy for Alcohol Use Disorder
Brief Title: Combination Therapy for Alcohol Use Disorder
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IRB00531545
Record Dates: First submitted 2025-11-18; First posted 2025-11-25 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Alcohol Use Disorder
Keywords: Glucagon-like peptide 1; Naltrexone; Alcohol Use Disorder; Addiction
MeSH Terms: conditions — Alcoholism; Behavior, Addictive | interventions — Naltrexone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Placebo+Placebo (Placebo Comparator): Placebo+Placebo
  Interventions: Drug: Placebo
- Placebo+GLP-1 (Experimental): Placebo+GLP-1
  Interventions: Drug: Placebo; Drug: Glucagon-Like Peptide-1 Agonist (GLP-1)
- GLP-1+Naltrexone (Experimental): GLP-1+Naltrexone
  Interventions: Drug: Glucagon-Like Peptide-1 Agonist (GLP-1); Drug: Naltrexone (oral tablets)

INTERVENTIONS:
Drug: Placebo — Over-encapsulated non-active microcrystalline cellulose
  Arms: Placebo+GLP-1; Placebo+Placebo
Drug: Glucagon-Like Peptide-1 Agonist (GLP-1) — Over-encapsulated Glucagon-Like Peptide-1 Agonist (GLP-1) oral tablets
  Arms: GLP-1+Naltrexone; Placebo+GLP-1
Drug: Naltrexone (oral tablets) — Over-encapsulated Naltrexone (oral tablets)
  Arms: GLP-1+Naltrexone

SUMMARY:
This human laboratory study will collect preliminary safety and efficacy data from a sample of participants enrolled in a 4-week in-patient treatment program for alcohol use disorder.

DETAILED DESCRIPTION:
Approximately 29 million persons in the United States aged 12 and older experienced a form of Alcohol Use Disorder (AUD) in 2023. Currently, only three pharmacotherapies are FDA-approved to treat AUD: acamprosate, naltrexone, and disulfiram. As monotherapies, these have shown moderate efficacy in reducing alcohol consumption and increasing abstinence. There is some evidence that therapeutic effects can be enhanced when combined with other medications. Recently, emerging preclinical evidence suggests that endogenous GLP-1 signaling plays a role in alcohol-mediated behaviors. Further, growing clinical data suggest that GLP-1 agonists (e.g., Wegovy, Rybelsus, Mounjaro) may be effective for the treatment of AUD. Studies evaluating the efficacy of GLP-1 agonists in combination with FDA-approved medications for AUD have yet to be conducted. The investigators hypothesize that combining a GLP-1 agonist and naltrexone may be more effective for reducing dimensions of AUD than naltrexone alone. The goal of this study is to collect preliminary safety and efficacy data from a sample of participants enrolled in a 4-week in-patient treatment program for AUD. Following one week of in-patient enrollment, participants will be randomized to one of three conditions in a double dummy design: placebo + placebo, GLP-1 + placebo, or GLP-1 + naltrexone. All study medications will be administered orally. Participants randomized to active GLP-1 conditions will receive 3 mg during study week 1 and can increase to 7 mg during week 2. Participants will attend study visits in a 14-day period to complete assessments of alcohol craving, alcohol demand, anhedonia, eating behaviors, and subjective effects. Participants will also provide vitals and biosamples to evaluate health outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Aged 21-65 years old
* Enrolled at Ashley Addiction Treatment center at least one week prior to beginning study participation.
* Meet the Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition, Text Revision (DSM-5-TR) criteria for Alcohol Use Disorder
* Willing to comply with the study protocol

Exclusion Criteria:

* Score 9 or greater on the Clinical Institute Withdrawal Assessment for Alcohol-Revised (CIWA-Ar) at randomization
* Currently pregnant, breastfeeding
* Unwilling to use contraceptives (e.g., condoms and/or hormonal birth control)
* Meet criteria for another substance use disorder other than AUD, Tobacco Use Disorder, or Caffeine use disorder
* History of pancreatitis
* History or current diagnosis of gallbladder disease, hepatic disease, renal disease, hyperparathyroidism, or any physical health condition that would be contraindicated with GLP-1 agonists or naltrexone.
* Unmanaged diabetes diagnosis or history or current diagnosis of diabetic retinopathy
* Levels of amylase, lipase, aspartate aminotransferase (AST), and/or alanine transferase (ALT) greater than 2x upper limit of normal
* Personal or family history of medullary thyroid carcinoma given FDA box warning for semaglutide
* Diagnosis of cancer within past 5 years
* History of multiple endocrine neoplasia syndrome type 2 (MEN2)
* Currently taking any medications contraindicated with GLP-1 agonists and/or naltrexone.
* BMI <18.5
* Current elevated suicide risk as assessed by clinic staff or the Columbia Suicide Severity Rating Scale (C-SSRS)
* Any other medical or psychological condition that is judged by the investigators to impede ability to safely complete study requirements.
* Legal problems or living situation judged by the investigators as a factor that could interfere with study completion (e.g., impending jail time).
* Allergies to semaglutide and/or naltrexone
* Use of opioids within the past 10 days as indicated by self-report or a positive urine drug screen
* Prescribed or taking the following medications in the past four weeks:
* The following medications will be prohibited during study participation due to interactions with semaglutide: other GLP-1 agonists (e.g. Exenatide, liraglutide, dulaglutide), insulin, insulin-secreting medications (e.g. sulfonylureas, meglitinides), tirzepetide, dipeptidyl peptidase-4 (DPP-4) inhibitors (e.g. sitagliptin, saxagliptin, linagliptin, alogliptin, evogliptin, and gemigliptin).
* The following medications will be prohibited during study participation due to interactions with naltrexone: bremelanotide, peripherally-acting mu-opioid receptor antagonists (e.g. methylnaltrexone, naldemedine), and opioid agonist medications.

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2026-03 (Estimated); Primary Completion 2028-03 (Estimated); Study Completion 2028-06 (Estimated)

PRIMARY OUTCOMES:
Participant-reported Adverse Events | 14 days
  Participant-reported adverse events during the course of the trial

CONTACTS AND LOCATIONS:
Overall Officials: Andrew S. Huhn, Ph.D., Principal Investigator — Johns Hopkins University
Locations (1):
- Ashley Addiction Treatment, Havre de Grace, Maryland, United States

IPD SHARING:
Plan to Share IPD: No
Data may be shared upon request.